CLINICAL TRIAL: NCT05348369
Title: The Relationship of Relative Corneal Refractive Power Shift and Axial Length in Adolescents With Orthokeratology Lens
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022020
Record Dates: First submitted 2022-04-20; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Myopia; Orthokeratology
Keywords: Myopia; Orthokeratology; Axial length
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Orthokeratology lens is an effective method for myopia control. This study analyzed the relationship between the relative corneal refractive power shift and change of axial length in adolescents with orthokeratology lens.

DETAILED DESCRIPTION:
Orthokeratology lens is an effective method for myopia control. This study aimed to investigate the relationship between the relative corneal refractive power shift and changes of axial length in adolescents with orthokeratology lens in 1 year. Other factors that may affect axial growth were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age from 8 to 15years
* spherical equivalent(SE) was range from -1.00D to -5.00D
* conform to the standard of wearing orthokeratology lens

Exclusion Criteria:

* ocular diseases and systemic diseases
* visual acuity was less than 20/20
* unable to follow visitors on time

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Myopia children with orthokeratology lens and complete follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of axial length | The change of baseline and 1years
  The axial length was measured by AL-scan, its expressed in mm

SECONDARY OUTCOMES:
Relative corneal refractive power shift(RCRPS) | up to 1 year
  The value of RCRPS was obtained and calculated from a corneal topography

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent SJ, Cho P, Chan KY, Fadel D, Ghorbani-Mojarrad N, Gonzalez-Meijome JM, Johnson L, Kang P, Michaud L, Simard P, Jones L. CLEAR - Orthokeratology. Cont Lens Anterior Eye. 2021 Apr;44(2):240-269. doi: 10.1016/j.clae.2021.02.003. Epub 2021 Mar 25. PMID 33775379
- [Background] Guo B, Cheung SW, Kojima R, Cho P. One-year results of the Variation of Orthokeratology Lens Treatment Zone (VOLTZ) Study: a prospective randomised clinical trial. Ophthalmic Physiol Opt. 2021 Jul;41(4):702-714. doi: 10.1111/opo.12834. Epub 2021 May 15. PMID 33991112